CLINICAL TRIAL: NCT02804542
Title: Pre-operative Fascia Iliaca Blocks and Opioid Requirements in Hip Fracture Patients
Brief Title: Fascia Iliaca Blocks and Pre-operative Opioid Requirements in Hip Fracture Patients
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Collaborators: Grand Rapids Medical Education Partners (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-160
Record Dates: First submitted 2016-06-01; First posted 2016-06-17 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hip Fracture
Keywords: fascia iliaca blocks
MeSH Terms: conditions — Hip Fractures | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fascia Iliaca Block Cohort: Prospective patients receiving fascia iliaca blocks A prospective Observational study of Hip fracture patients that are offered fascia iliaca blocks as standard of care in the ED.
  Interventions: Other: Observational
- Retrospective Control Cohort: No fascia iliaca block performed A retrospective review will be done of hip fracture patients that did not receive fascia iliaca blocks (before fascia iliaca blocks being offered in the ED as standard of care).
  Interventions: Other: Retrospective review

INTERVENTIONS:
Other: Observational
  Groups: Fascia Iliaca Block Cohort
Other: Retrospective review
  Groups: Retrospective Control Cohort

SUMMARY:
The purpose of this study is to determine if non-continuous local anesthetic fascia iliaca blocks performed in the emergency department are effective for preoperative analgesia in hip fracture patients. Investigators hypothesize that patients with these blocks will have lower opioid requirements than patients in a historical group in whom blocks were not performed.

ELIGIBILITY:
Inclusion Criteria:

* low energy femoral neck and pertrochanteric-type hip fractures
* age 65+
* intact cognition upon admission and ability to provide written informed consent

Exclusion Criteria:

* pathologic fractures (tumor)
* high energy fractures
* concomitant fractures besides hip fractures
* chronic home opioid exposure prior to hospitalization
* moderate to severe dementia
* pre-fracture hospitalization
* time from arrival to block >6 hours
* time from arrival to OR <6 hours or >48 hours

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients >65 years of age presenting to Spectrum Health Butterworth hospital with low-energy hip fractures (displaced and non-displaced femoral neck, pertrochanteric-type including subtrochanteric extension) will be screened for the study.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Total Pre-op IV Morphine Equivalents (TIVME) | From Date of admission until date of surgery, approximately 48 hours
  IV morphine equivalent dosing pre-operatively

SECONDARY OUTCOMES:
Mean Pre-op Pain Score | From Date of admission until date of surgery, approximately 48 hours
  Mean patient-reported pain score
Length of Hospital Stay (LOS) | Through study completion, approximately 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Flannigan, MD, Principal Investigator — ECS

IPD SHARING:
Plan to Share IPD: No